CLINICAL TRIAL: NCT06702579
Title: Qualitative Study on Home Monitoring of Hemostasis in Anticoagulant Treatment and Hemophilia a
Brief Title: Home Monitoring in Hemophilia a
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: HEMSTOL85
Record Dates: First submitted 2024-11-12; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Hemophilia a; Anticoagulant Therapy; Monitoring; Point of Care Testing; Qualitative Research
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patients receiving anticoagulation therapy: Adult patients on anticoagulation therapy who perform INR self-testing at home.
- Hemophilia A: Patients over 12 years old with congenital hemophilia A receiving prophylactic therapy.
- Healthcare professionals: Hematologists, hemophilia nurses, pharmacists or other healthcare providers currently involved in the care for patients with hemophilia.

SUMMARY:
Rationale: A novel point-of-care device capable of measuring factor VIII (FVIII) activity and thrombin generation (TG) is currently under development. Utilization of this device in a home situation could potentially transform hemophilia care and improve patients' autonomy.

Objective: To explore the potential consequences of home monitoring of hemostatic parameters in patients with hemophilia A

Study design: Cross-sectional observational study consisting of semi-structured interviews and focus groups

Study population: Approximately 10 patients treated with vitamin K antagonists engaging in self-monitoring of coagulation at home and approximately 20 patients with hemophilia A.

Main study parameters/endpoints: The main outcome of this study is to assess series of interrelated themes related to the unmet needs of hemophilia patients and the envisioned potential consequences of home monitoring on these unmet needs.

Secondary outcomes include: identifying key features of a home monitoring platform to be used in hemophilia care, describing the experienced consequences of implementing home self-monitoring in anticoagulation treatment, assessing the current experiences of patients with self-monitoring, and providing an overview of the burdens and unmet needs experienced by patients with hemophilia with current hemophilia care.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The risk associated with participation in this study is negligible. Minor patients will be included in this study only if informed consent is given by both the patient and his/her caregiver (in patients between 12-16 years old). Gathering the insights of caregivers of minor patients on the current care for hemophilia and potential consequences of home self-monitoring is vital, as their experiences and needs might differ significantly from older patients. Participating in this study does not entail direct benefits. However, patients who participate can contribute to the development of future monitoring systems, which have the potential to alleviate the current burden of their disease and treatment.

ELIGIBILITY:
Patients treated with vitamin K antagonists Inclusion criteria

* Aged > 16 years
* Patient using vitamin K antagonist for any indication
* Registered at the "Trombosezorg dichterbij"
* Self-testing INR at home for > 3 months
* A history of monitoring INR at a care facility (not self-testing)
* Signed informed consent form
* Able to speak and understand Dutch or English without a translator

Exclusion criteria

• Unwilling to consent with the study or with audio recording

Hemophilia A patients Inclusion criteria

* Diagnosis of congenital hemophilia A, with or without inhibitors
* Receiving prophylactic treatment
* Patients aged ≥ 12 years or caregivers of patients aged < 12 years old
* Signed informed consent form
* Able to speak and understand Dutch or English without a translator Exclusion criteria
* No diagnosis of congenital hemophilia A
* Unwilling to consent with the study or with audio recording

Hemophilia healthcare professionals Inclusion criteria

* Hematologist, hemophilia nurse, pharmacist or healthcare provider currently involved in the care for patients with hemophilia
* At least > 3 years clinical experience in hemophilia care
* Signed informed consent form
* Able to speak and understand Dutch or English without a translator

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The exact sample size for this study is not predetermined. Instead, patients will be selected using purposeful sampling methodology until theoretical saturation is achieved. Maximum variation in age, severity of hemophilia and received treatment will be pursued.
  Three cases are included in the study:
  1. Patients registered at the "Trombosezorg dichterbij", treated with a vitamin K antagonist for any indication, currently engaging in self-testing INR at home
  2. Patients and caregivers of patients with hemophilia A, who require prophylactic therapy with a factor VIII concentrate. Hemophilia patients will be sampled from the patients receiving care from the Hemophilia Treatment Center Nijmegen Eindhoven Maastricht. If insufficient patients can be included from this population to achieve data saturation, additional patients will be sampled via the patient society
  3. HCPs involved in the treatment of hemophilia patients and technical experts to provide additional context.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Semi structured interviews - identified themes on the potential impact of home monitoring in the care for patients with hemophilia A | At enrollment
  Interrelated themes describing the current experiences and envisioned impact of home monitoring in hemophilia A, derived from analysis of semi-structured qualitative interviews (thematic analysis as described by Braun and Clarke (2006))

SECONDARY OUTCOMES:
Semi-structured interview - Themes describing the current experienced burdens and unmet needs for hemophilia A patients requiring prophylactic therapy | At enrollment
  Interrelated themes describing current experienced burdens and unmet needs for hemophilia A patients requiring prophylactic therapy, derived from analysis of semi-structured qualitative interviews (thematic analysis as described by Braun and Clarke (2006))
Semi-structured interviews - Identified themes on the current experiences of patients receiving anticoagulation with coagulation home monitoring | At enrollment
  Interrelated themes describing the experiences of patients receiving anticoagulation with coagulation home monitoring, derived from analysis of semi-structured qualitative interviews (thematic analysis as described by Braun and Clarke (2006))
Focus groups - Identified themes on healthcare providers' expectations regarding home monitoring in hemophilia A | At enrollment
  Interrelated themes describing the expectations of healthcare providers on the impact of home monitoring in hemophilia A, derived from analysis of semi-structured qualitative interviews (thematic analysis as described by Braun and Clarke (2006))

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No